CLINICAL TRIAL: NCT05184465
Title: Comparison of the Efficacy of 0.5% Bupivacaine, 0.5% Levobupivacaine, and 0.5% Hyperbaric Bupivacaine in Equal Volumes for Spinal Anesthesia in Lower Limb Surgeries
Brief Title: Comparison of the Efficacy of 0.5% Bupivacaine, 0.5% Levobupivacaine, and 0.5% Hyperbaric Bupivacaine
Acronym: BvsLBvsHB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mogilev Regional Clinical Hospital (Other Government)
Responsible Party: Principal Investigator, Valery Piacherski, Ph.D., Chief of the Department of Anesthesiology and Intensive Care, Mogilev Regional Clinical Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 28.01.2017
Record Dates: First submitted 2021-12-01; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Anesthesia, Spinal
Keywords: Bupivacaine; Levobupivacaine; Hyperbaric bupivacaine; Anesthesia Spinal; Аnesthetics Local
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bupivacaine (Experimental): Spinal anesthesia was administered to the patients for anesthetic support of the surgical intervention.Intrathecal injections were performed with a 24G or 25G "Pencil point" needle in the L3-L4 interval. Spinal puncture was performed while the patient was sitting on the table.Spinal anesthesia was performed with 3 ml of 0.5% bupivacaine. Then the patient was placed on his back.Surgery was allowed to start after 40 minutes if the upper level of the sensory block reached the Th10 segment.
  Interventions: Procedure: spinal anesthesia
- Levobupivacaine (Experimental): Spinal anesthesia was administered to the patients for anesthetic support of the surgical intervention.Intrathecal injections were performed with a 24G or 25G "Pencil point" needle in the L3-L4 interval. Spinal puncture was performed while the patient was sitting on the table.Spinal anesthesia was performed with 3 ml of 0.5% Levobupivacaine. Then the patient was placed on his back.Surgery was allowed to start after 40 minutes if the upper level of the sensory block reached the Th10 segment.
  Interventions: Procedure: spinal anesthesia
- Hyperbaric bupivacaine (Experimental): Spinal anesthesia was administered to the patients for anesthetic support of the surgical intervention.Intrathecal injections were performed with a 24G or 25G "Pencil point" needle in the L3-L4 interval. Spinal puncture was performed while the patient was sitting on the table.Spinal anesthesia was performed with 3 ml of 0.5% Hyperbaric bupivacaine. Then the patient was placed on his back.Surgery was allowed to start after 40 minutes if the upper level of the sensory block reached the Th10 segment.
  Interventions: Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — The anesthesiologist, who was not involved in the study, prepared the anesthetic solution immediately before the injection.
  Intrathecal injections were performed with a 24G or 25G "Pencil point" needle in the L3-L4 interval. Spinal puncture was performed while the patient was sitting on the table. Then the patient was placed on his back.

SUMMARY:
About 15 million spinal anesthesia procedures are performed worldwide each year. In the daily practice of the anesthesiologist for intrathecal use there are various local anesthetics such as bupivacaine, hyperbaric solution of bupivacaine, ropivacaine and levobupivacaine. From 1946 to 2017, only 16 studies comparing the clinical efficacy of isobaric and hyperbaric bupivacaine in nonpregnant patients have been conducted according to various databases. The small sample size and high heterogeneity of these results suggest that all results should be treated with caution. And, there is no conclusive evidence in favor of isobaric or hyperbaric bupivacaine regarding efficacy or side effects in the general surgical population.

The literature describes such advantages of levobupivacaine as less cardiotoxicity, longer period of analgesia, more pronounced activity against sensory fibers than against motor fibers. In some studies it has been shown that levobupivacaine is equal to isobaric bupivacaine in efficacy. The efficacy of hyperbaric levobupivacaine equivalent to hyperbaric bupivacaine when administered intrathecally has also been shown on volunteers.

However, in the literature there are different data on clinical efficacy of levobupivakin in comparison with ropivacaine and levobupivacaine. So during operations on extremities out of 20 patients surgical anesthesia developed in 18 patients. Fattorini F. et al. D in their study stated the same effectiveness of bupivacaine and levobupivacaine, but when using levobupivacaine in one patient general anesthesia was used due to insufficient spinal anesthesia. Other studies also reported similar efficacy of the two drugs, but surgical satisfaction with intraoperative anesthesia was 92.9% for bupivacaine and 83.9% for levobupivacaine for knee arthoroscopy.

In their study, P Gautier et al. noted significantly lower efficacy of levobupivacaine in caesarean section compared to bupivacaine and ropivacaine for intrathecal use: 80% vs. 90% and 87%, respectively.

According to Heng Sia et al. there is no clear evidence of the advantage of hyperbaric bupivacaine over isobaric bupivacaine for spinal anesthesia for cesarean section. The authors also noted that adequate randomized clinical trials with clear definitions, criteria and methodology for evaluating the transition to general anesthesia, requirements for additional analgesia, nausea, vomiting and sensory testing are needed.

There is no clear practical guide to help anesthesiologists make informed decisions about the use of some form of intrathecal bupivacaine in non-cesarean surgery. Carefully designed, adequately conducted studies can provide further results that will contribute to sound clinical decision making.

Given the above, the aim of the study is to compare the effectiveness of spinal anesthesia (SA) performed with 0.5% isobaric bupivacaine solution, 0.5% levobupivacaine solution and 0.5% hyperbaric bupivacaine solution in equivalent volumes in lower limb surgeries.

DETAILED DESCRIPTION:
111patients who underwent surgical intervention on the hip, thigh, and knee joints were included in the study.

Criteria for inclusion of patients in the study: indications for surgical intervention on the hip, thigh, and knee joints. Anesthesiological support was required; a written informed consent was obtained from patients to participate in the clinical trial and a written informed consent of the patient about the type of anesthesia and possible complications of regional anesthesia was available. After obtaining informed consent, patients were randomized into groups using a random number generator (numbers in envelopes). The random assignment sequence was created by an anesthesiologist not involved in the study.

Exclusion criteria: patient refusal to use the proposed type of anesthesia, age <18 years, body mass index not > 39, physical status according to ASA 1-3, history of allergic reactions to the drugs used, coagulopathy, infectious skin lesions in the injection area, neurological or neuromuscular diseases, severe liver disease or renal failure, inability to cooperate with the patient.

Spinal anesthesia was administered to the patients for anesthetic support of the surgical intervention. Patients were randomly allocated into three groups: in group 1 (1B) spinal anesthesia was performed with 3 ml of 0.5% bupivacaine(n=37); in group 2 (2L) spinal anesthesia was performed with 3 ml of 0.5% levobupivacaine (n=37); in group 3 (3H) 3 ml of 0.5% hyperbaric bupivacaine solution (n=37) was used for subarachnoid injection. The anesthesiologist, who was not involved in the study, prepared the anesthetic solution immediately before the injection.

Intrathecal injections were performed with a 24G or 25G "Pencil point" needle in the L3-L4 interval. Spinal puncture was performed while the patient was sitting on the table. Then the patient was placed on his back.

Solutions for spinal anesthesia were prepared by an anesthesiologist who was not involved in the anesthesia. Spinal anesthesia was performed by an anesthesiologist with many years of experience, who performs 10-15 spinal anesthesias per week.

The peripheral vein was catheterized on the operating table before anesthesia. SPO2, ECG, HR, thermometry, and nBP were monitored during anesthesia and surgery.

Surgery was allowed to start after 40 minutes if the upper level of the sensory block reached the Th10 segment.

The criterion for assessing the effectiveness of anesthesia was the need to switch to another type of anesthesia (criterion-no anesthesia), or the need for additional use of narcotic analgesics or local anesthesia during surgery (criterion-reporting of painful feelings during the operation).

The block was evaluated by an anesthesiologist who was not involved in the study. Sensory block quality was recorded on both sides along the midclavicular line, assessing changes in needle prick sensation. Skin sensitivity was assessed every 2 minutes for 40 minutes. The following scale was used to assess sensory block, where: "++" - complete sensory block (anesthesia); "+" - not complete sensory block, the patient could not differentiate the type of stimulus; "˗" - skin sensitivity preserved to the full extent.

The development of motor block was assessed using the Bromage scale (0-3) for 40 minutes. End of motor block was defined as the appearance of the first movements in the lower extremities (within 24 hours).

The duration of postoperative analgesia was assessed by interviewing the patient in the postoperative period (within 24 hours). The duration of analgesia was assessed in the postoperative period every 30 minutes. Pain sensations were assessed by visual analog scale (VAS) from 0 cm (no pain) to 10 cm (unbearable pain). The end of analgesia was considered the moment when the patient noted the onset of pain (1-2 points). If painful sensations appeared in the postoperative wound area (1-2 points),the investigators injected intramuscularly 2 %-1 ml of Promedol for postoperative analgesia. The duration of analgesia was assessed by an independent anesthesiologist, who was not involved in the study.

For the additional intraoperative analgesia criterion, the null hypothesis implies that the degree of success in the compared groups (for each local anesthetic) is the same ( p >0.05). If the null hypothesis should be rejected after a statistical test ( p < 0.05), it is concluded that one of the groups is superior to the others on this indicator. The sample size was calculated for a confidence level of 99% and statistical power of 99% and a type 1 error of 0.01 (taking into account the effectiveness of performing spinal anesthesia with bupivacaine 0.5% in orthopedics at our institution). The estimated sample size for each group was 7 patients. Considering previous studies in this area, where the sample size ranged from 29 to 40 patients, the investigators included an additional 30 patients in each group to increase validity (total 37 patients in each group).

Statistical processing of the obtained data was performed using Statistica 7.0 software. The data were presented as median and quartiles (25th% and 75th%) and also as mean and standard deviation. Differences between the groups were considered statistically significant at p<0.05. The primary endpoint was the need to switch to another type of anesthesia or the need for additional narcotic analgesics or local anesthesia either initially or during surgery. The frequencies of the binary feature in the two unrelated (independent) groups were compared by analysis of a contingency table (2×2). Classic Pearson's X2 test (Chi-square) was used; Fisher exact p test was applied in the presence of values of the phenomena of 5 and less. Differences between the groups were considered statistically significant at p<0.05. 95% CI for categorical data calculated using Wald's method.

Secondary endpoints: time of sensory and motor block development, duration of postoperative analgesia and motor block. The groups were compared using nonparametric Mann-Whitney test. Differences between the groups were considered statistically significant at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* indications for surgical intervention on the hip, thigh, and knee joints

Exclusion Criteria:

* patient refusal to use the proposed type of anesthesia,
* age <18 years,
* body mass index not > 39,
* physical status according to ASA 1-3,
* history of allergic reactions to the drugs used,
* coagulopathy,
* infectious skin lesions in the injection area,
* neurological or neuromuscular diseases,
* severe liver disease or renal failure,
* inability to cooperate with the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
Effectiveness of anesthesia | Intraoperative
  The criterion for assessing the effectiveness of anesthesia was the need to switch to another type of anesthesia (criterion-no anesthesia), or the need for additional use of narcotic analgesics or local anesthesia during surgery (criterion-reporting of painful feelings during the operation).

SECONDARY OUTCOMES:
Complete sensory block | Skin sensitivity was assessed every 2 minutes for 40 minutes
  The following scale was used to assess sensory block, where: "++" - complete sensory block (anesthesia); "+" - not complete sensory block, the patient could not differentiate the type of stimulus; "˗" - skin sensitivity preserved to the full extent.
Complete motor block | Motor block was assessed every 2 minutes for 40 minutes
  The development of motor block was assessed using the Bromage scale (0-3) for 40 minutes.
Time to develop a complete sensory block, (min) | Skin sensitivity was assessed every 2 minutes for 40 minutes
  The following scale was used to assess sensory block, where: "++" - complete sensory block (anesthesia); "+" - not complete sensory block, the patient could not differentiate the type of stimulus; "˗" - skin sensitivity preserved to the full extent.
Time of development of the full motor block, (min) | Motor block was assessed every 2 minutes for 40 minutes
  The development of motor block was assessed using the Bromage scale (0-3) for 40 minutes.
Duration of analgesia, (min) | Postoperative period (within 24 hours)
  The duration of postoperative analgesia was assessed by interviewing the patient in the postoperative period (within 24 hours). The duration of analgesia was assessed in the postoperative period every 30 minutes. Pain sensations were assessed by visual analog scale (VAS) from 0 cm (no pain) to 10 cm (unbearable pain). The end of analgesia was considered the moment when the patient noted the onset of pain (1-2 points). If painful sensations appeared in the postoperative wound area (1-2 points), we injected intramuscularly 2 %-1 ml of Promedol for postoperative analgesia. The duration of analgesia was assessed by an independent anesthesiologist, who was not involved in the study.
Duration of motor block, (min) | Postoperative period (within 24 hours)
  End of motor block was defined as the appearance of the first movements in the lower extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Valery Piacherski, Principal Investigator — Mogilev Regional Clinical Hospital
Locations (1):
- Mogilev Regional Clinical Hospital, Mogilev, Belarus

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data can be provided after the publication of the results of our study in a scientific medical journal.With the condition of reference to the authors of this study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual participant data can be provided after the publication of the results of our study in a scientific medical journal.
Access Criteria: Apply to the e-mail address to the authors: pechersky.v@yandex.ru

REFERENCES:
- [Background] Uppal V, Retter S, Shanthanna H, Prabhakar C, McKeen DM. Hyperbaric Versus Isobaric Bupivacaine for Spinal Anesthesia: Systematic Review and Meta-analysis for Adult Patients Undergoing Noncesarean Delivery Surgery. Anesth Analg. 2017 Nov;125(5):1627-1637. doi: 10.1213/ANE.0000000000002254. PMID 28708665
- [Background] Foster RH, Markham A. Levobupivacaine: a review of its pharmacology and use as a local anaesthetic. Drugs. 2000 Mar;59(3):551-79. doi: 10.2165/00003495-200059030-00013. PMID 10776835
- [Background] del-Rio-Vellosillo M, Garcia-Medina JJ, Abengochea-Cotaina A, Pinazo-Duran MD, Barbera-Alacreu M. Spinal anesthesia for knee arthroscopy using isobaric bupivacaine and levobupivacaine: anesthetic and neuroophthalmological assessment. Biomed Res Int. 2014;2014:349034. doi: 10.1155/2014/349034. Epub 2014 Feb 20. PMID 24701571
- [Background] Glaser C, Marhofer P, Zimpfer G, Heinz MT, Sitzwohl C, Kapral S, Schindler I. Levobupivacaine versus racemic bupivacaine for spinal anesthesia. Anesth Analg. 2002 Jan;94(1):194-8, table of contents. doi: 10.1097/00000539-200201000-00037. PMID 11772827
- [Background] Alley EA, Kopacz DJ, McDonald SB, Liu SS. Hyperbaric spinal levobupivacaine: a comparison to racemic bupivacaine in volunteers. Anesth Analg. 2002 Jan;94(1):188-93, table of contents. doi: 10.1097/00000539-200201000-00036. PMID 11772826
- [Background] Burke D, Kennedy S, Bannister J. Spinal anesthesia with 0.5% S(-)-bupivacaine for elective lower limb surgery. Reg Anesth Pain Med. 1999 Nov-Dec;24(6):519-23. doi: 10.1016/s1098-7339(99)90042-1. PMID 10588555
- [Background] Fattorini F, Ricci Z, Rocco A, Romano R, Pascarella MA, Pinto G. Levobupivacaine versus racemic bupivacaine for spinal anaesthesia in orthopaedic major surgery. Minerva Anestesiol. 2006 Jul-Aug;72(7-8):637-44. English, Italian. PMID 16865082
- [Background] Gautier P, De Kock M, Huberty L, Demir T, Izydorczic M, Vanderick B. Comparison of the effects of intrathecal ropivacaine, levobupivacaine, and bupivacaine for Caesarean section. Br J Anaesth. 2003 Nov;91(5):684-9. doi: 10.1093/bja/aeg251. PMID 14570791
- [Background] Heng Sia AT, Tan KH, Sng BL, Lim Y, Chan ESY, Siddiqui FJ. Hyperbaric versus plain bupivacaine for spinal anesthesia for cesarean delivery. Anesth Analg. 2015 Jan;120(1):132-140. doi: 10.1213/ANE.0000000000000443. PMID 25625258
- [Background] Sng BL, Siddiqui FJ, Leong WL, Assam PN, Chan ES, Tan KH, Sia AT. Hyperbaric versus isobaric bupivacaine for spinal anaesthesia for caesarean section. Cochrane Database Syst Rev. 2016 Sep 15;9(9):CD005143. doi: 10.1002/14651858.CD005143.pub3. PMID 27629425
- [Background] Vernhiet J, Cheruy D, Maindivide J, Vabre M, Clement C, Dartigues JF. [Spinal anesthesia with bupivacaine. Comparative study of 2 hyperbaric and isobaric solutions]. Ann Fr Anesth Reanim. 1984;3(4):252-5. doi: 10.1016/s0750-7658(84)80115-x. French. PMID 6476498
- [Background] Singh A, Gupta A, Datta PK, Pandey M. Intrathecal levobupivacaine versus bupivacaine for inguinal hernia surgery: a randomized controlled trial. Korean J Anesthesiol. 2018 Jun;71(3):220-225. doi: 10.4097/kja.d.18.27191. Epub 2018 Apr 24. PMID 29684982
- [Derived] Piacherski V, Muzyka L. Comparison of the efficacy of 0.5% isobaric bupivacaine, 0.5% levobupivacaine, and 0.5% hyperbaric bupivacaine for spinal anesthesia in lower limb surgeries. Sci Rep. 2023 Feb 15;13(1):2736. doi: 10.1038/s41598-023-29711-9. PMID 36792639